CLINICAL TRIAL: NCT06458101
Title: Efficacy and Safety of Ureteroscopic Lithotripsy (Including Flexible Ureteroscopy) Without Indwelling Urinary Catheter: a Multicenter, Randomized, Controlled Study
Brief Title: Efficacy and Safety of Ureteroscopic Lithotripsy (Including Flexible Ureteroscopy) Without Indwelling Urinary Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yi Shao, Director, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIT2024-050
Record Dates: First submitted 2024-06-03; First posted 2024-06-13 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Urolithiasis; Catheter-related Bladder Discomfort
MeSH Terms: conditions — Urolithiasis | interventions — Ureteroscopy; Lithotripsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Ureteroscopy (including flexible endoscope) lithotripsy with indwelling urinary catheter (Active Comparator): Ureteroscopy (including flexible endoscope) lithotripsy with indwelling urinary catheter
  Interventions: Procedure: Ureteroscopy (including flexible endoscope) lithotripsy with indwelling urinary catheter
- Group 2: Ureteroscopy (including flexible endoscope) lithotripsy without indwelling urinary catheter (Experimental): Ureteroscopy (including flexible endoscope) lithotripsy without indwelling urinary catheter
  Interventions: Procedure: Ureteroscopy (including flexible endoscope) lithotripsy without indwelling urinary catheter

INTERVENTIONS:
Procedure: Ureteroscopy (including flexible endoscope) lithotripsy without indwelling urinary catheter — Ureteroscopy (including flexible endoscope) lithotripsy without indwelling urinary catheter
  Arms: Group 2: Ureteroscopy (including flexible endoscope) lithotripsy without indwelling urinary catheter
Procedure: Ureteroscopy (including flexible endoscope) lithotripsy with indwelling urinary catheter — Ureteroscopy (including flexible endoscope) lithotripsy with indwelling urinary catheter
  Arms: Group 1: Ureteroscopy (including flexible endoscope) lithotripsy with indwelling urinary catheter

SUMMARY:
A prospective, multicenter, randomized, controlled clinical trial was conducted to compare the efficacy and safety of non-indwelling catheter and indwelling catheter in relieving postoperative catheter-related complications after ureteroscopic lithotripsy. By comparing the pain score and urination urgency score (PPIUS) of patients after ureteroscopic lithotripsy (including flexible ureteroscopy) lithotripsy to provide a reliable scientific basis for indwelling catheter after ureteroscopic lithotripsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with upper urinary tract calculi undergoing rigid ureteroscopic and soft ureteroscopic lithotripsy;
* Normal renal function;
* Aged between 18 and 70 years old
* Complete the operation under general anesthesia

Exclusion Criteria:

* Solitary kidney;
* Previous history of renal transplantation or urinary diversion;
* Congenital malformation of urinary system;
* Abnormal coagulation mechanism due to blood system diseases, liver diseases, etc.
* Severe heart or lung disease, Malignant tumor and immunodeficiency state
* Urethral stricture
* Neurogenic bladder
* Operation under epidural anesthesia or spinal anesthesia
* Large amount of bleeding during operation should be observed by indwelling catheter to observe urine color
* High risk factors such as large amount of pus fur should be observed during operation.
* Urethral injury during operation leads to false passage
* Operation time is more than 90 minutes. Higher risk of bleeding or infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Pain score | 4 hours after surgery and 2 hours after catheter removal (same time points for non-indwelling catheters)
  pain scoring will be measured by VAS scale. There are 10 scales, with "0" and "10" at both ends. 0 indicates no pain and 10 represents the most severe pain that is unbearable.
Urinary urgency score | 4 hours after surgery and 2 hours after catheter removal (same time points for non-indwelling catheters)
  urinary urgency score will be measured by PPIUS scale. 0 No urgency
  1. Mild urgency
  2. Moderate urgency
  3. Severe urgency
  4. Urge incontinence

SECONDARY OUTCOMES:
Painful Memory | 1 month after surgery
  Painful memory will be measured by SUDS scale. 100: Unbearably upset to the point that you cannot function and may be on the verge of a breakdown 90: Extremely anxious and desperate; helpless and unable to handle it 80: Worried and panicky; losing focus and feeling anxious in your body 70: Discomfort dominates your thoughts and you struggle to function normally 60: Moderate to strong levels of discomfort 50: Upset and uncomfortable; still functional 40: Mild to moderate anxiety and worry 30: Worried or upset; still able to function 20: A little bit sad or distressed 10: No distress; alert and focused 0: Peaceful and complete calm
Operation time | The end of operation
  Operation time
blood routine | Before surgery and 4 hours after surgery
  To calculate the change of haemoglobin

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
After the trial is completed, it is shared on the network platform: China Clinical trial Registration Center; website: http://www.chictr.org.cn
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After the trial is completed,
URL: http://www.chictr.org.cn